CLINICAL TRIAL: NCT03874871
Title: Function Preserving Gastrectomy for T1/2 Gastric Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); Peking Union Medical College Hospital (Other); Beijing Friendship Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Beijing Hospital (Other Government); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Ziyu Li, MD, Principal Investigator, Clinical Professor, Peking University
Other Study IDs: 2018KT86
Record Dates: First submitted 2019-03-04; First posted 2019-03-14 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Gastric Cancer; Gastrostomy
Keywords: gastric cancer; function preserving gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Function preserving gastrectomy: After baseline evaluation, a multidisciplinary discussion will be performed for the patients to choose the proper gastrectomy. For patients indicated for function preserving gastrectomy (including pylorus preserving gastrectomy, proximal gastrectomy, partial gastrectomy), they will receive the function preserving gastrectomy. After the surgery, a close follow up is performed.
  Interventions: Procedure: Function preserving gastrectomy
- Standard gastrectomy: After baseline evaluation, a multidisciplinary discussion will be performed for the patients to choose the proper gastrectomy. For patients not indicated for function preserving gastrectomy, they will receive standard gastrectomy. After the surgery, a close follow up is performed.
  Interventions: Procedure: Standard gastrectomy

INTERVENTIONS:
Procedure: Function preserving gastrectomy — Function preserving gastrectomy include pylorus preserving gastrectomy, proximal gastrectomy, and partial gastrectomy.
  Groups: Function preserving gastrectomy
Procedure: Standard gastrectomy — Standard gastrectomy include distal gastrectomy and total gastrectomy with standard lymphadenectomy according to the Japanese gastric cancer treatment guideline.
  Groups: Standard gastrectomy

SUMMARY:
The real world based multi-cohorts study aims to evaluate the safety and effectiveness of function preserving gastrectomy including pylorus-preserving distal gastrectomy, proximal gastrectomy and wedge gastrectomy for T1 and T2 gastric cancer patients.

DETAILED DESCRIPTION:
Gastric cancer patients with clinical stage T1/2 will be screened for the study. For the patients enrolled, a multidisciplinary discussion will be performed to evaluate the proper gastrectomy for the patients and functional preserving gastrectomy will be considered for the indicated patients. For patients not proper for functional preserving gastrectomy, standard gastrectomies will be suggested. After surgery, a close follow up will be performed. During the study, a thorough data collection will be performed to evaluate the safety and effectiveness of functional preserving gastrectomy and recovery and postoperative function of remnant stomach.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance over 70%
* Histologically proven gastric or gastroesophageal joint adenocarcinoma with clinical stage T1-2N0-3M0
* No severe comorbidity with estimated survival less than 5 years

Exclusion Criteria:

* pregnancy
* Signs of distant metastases
* received chemotherapy, radiotherapy, immune therapy
* received gastrectomy
* other malignant tumors within 5 years except for cured skin cancer and cervical caner in situ.
* uncontrolled epilepsy, central nervus system disease or mental disease that affect the compliance of treatment and follow-up
* severe heart disease
* organ transplantation that needs immunosuppressor
* emergency surgery due to hemorrhage, perforation and ileus of gastric cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-advanced gastric cancer patients with the clinical stage cT1-2 that are indicated for gastrectomy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 30 days after surgery
  Pathologic R0 resection rate with negative proximal and distal margin based on the postoperative pathologic result.

SECONDARY OUTCOMES:
Extent of lymphadenectomy of different gastrectomy | 30 days after surgery
  resected lymph node number
Distribution of metastatic lymph node | 30 days after surgery
  metastatic lymph node number
postoperative morbidity | 30 days after surgery
  postoperative complication rate according to the clavien-dindo classification
postoperative mortality | 30 days after surgery
  postoperative death rate with 30 days
remnant stomach function | 3 years after surgery
  volume of remnant stomach
disease free survival | 3 years after surgery
  disease free survival after surgery
Quality of life after surgery | 3 years after surgery
  Quality of life evaluated by EORTC-STO22 by questionnaire
overall survival | 3 years after surgery
  overall survival after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ziyu Li, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No